CLINICAL TRIAL: NCT06137066
Title: The Effect of Green Coffee Extract With Alpha-lipoic Acid or Dihydroberberine on Blood Glucose Homeostasis in Healthy Adults
Brief Title: The Effect of Green Coffee Extract on Blood Glucose Homeostasis in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Chris McGlory, PhD (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Sponsor-Investigator, Dr. Chris McGlory, PhD, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 6039146
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Green Coffee Extract; Chlorogenic Acid; Alpha-Lipoic Acid; Dihydroberberine
MeSH Terms: interventions — dihydrodibutylstilbestrol

STUDY DESIGN:
Intervention Model Description: Four-arm study. All participants receive all acute nutritional interventions: placebo (microcrystalline cellulose with 5mg magnesium stearate and 5mg silicon dioxide), 200mg GCE +200mg ALA, 200mg GCE + 400mg ALA, 200mg GCE + 200mg dihydroberberine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Supplements will be coded as either 'A', 'B', 'C', or 'D'. A third-party researcher not involved in data collection will store the code key and only reveal the information after the data has been analyzed to maintain the double-blinded nature of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo supplement consisting of microcrystalline cellulose with 5mg magnesium stearate and 5mg silicon dioxide.
  Interventions: Dietary Supplement: Placebo
- 200mg GCE +200mg ALA (Experimental): 200mg green coffee extract +200mg alpha-lipoic acid
  Interventions: Dietary Supplement: 200mg GCE +200mg ALA
- 200mg GCE +400mg ALA (Experimental): 200mg green coffee extract +200mg alpha-lipoic acid
  Interventions: Dietary Supplement: 200mg GCE +400mg ALA
- 200mg GCE +200mg DHB (Experimental): 200mg green coffee extract + 200mg dihydroberberine
  Interventions: Dietary Supplement: 200mg GCE + 200mg DHB

INTERVENTIONS:
Dietary Supplement: 200mg GCE +200mg ALA — 200mg green coffee extract + 200mg alpha-lipoic acid
  Arms: 200mg GCE +200mg ALA
Dietary Supplement: 200mg GCE +400mg ALA — 200mg green coffee extract + 400mg alpha-lipoic acid
  Arms: 200mg GCE +400mg ALA
Dietary Supplement: 200mg GCE + 200mg DHB — 200mg green coffee extract + 200mg dihydroberberine
  Arms: 200mg GCE +200mg DHB
Dietary Supplement: Placebo — microcrystalline cellulose with 5 mg magnesium stearate and 5 mg silicon dioxide
  Arms: Placebo

SUMMARY:
Green coffee extract (GCE) supplementation has been shown to induce favourable health benefits on glucose metabolism and weight management. Previous literature suggests that the benefits of GCE are due to the high bioavailability of chlorogenic acid (CGA) which is known for its antioxidant and anti-inflammatory properties but is destroyed during the bean roasting process used to make coffee in Western societies. While some studies examining chronic and high-dose GCE supplementation (4-12 weeks) report beneficial effects on glucose handling and reductions in body mass following supplementation, comparably less is known about the effect of acute (single dose) GCE supplementation. The purpose of the current study is to determine the impact of acute supplementation of GCE on blood sugar levels following consumption of a carbohydrate drink in healthy adults. A secondary objective is to evaluate the effect of GCE on insulin levels, other measures of glucose metabolism, and appetite perceptions.

DETAILED DESCRIPTION:
Green coffee extract (GCE) supplementation has been shown to induce favourable benefits on glucose metabolism and weight management. These effects are attributed to its high chlorogenic acid (CGA) content, recognized for its anti-inflammatory properties. Chronic CGA supplementation (4-12 weeks) has been linked to reduced body mass, waist circumference, fasting glucose, and insulin resistance in both healthy adults and those with metabolic disease. Yet, comparably fewer studies have examined the effects of acute GCE supplementation and yielded inconsistent results, likely owing to variations in study design and participant selection, which limit our understanding of its acute effects.

Alpha-lipoic acid (ALA) is a cofactor of mitochondrial dehydrogenase complexes and a potent antioxidant that has been implicated in glucose metabolism. ALA increases the translocation of glucose transporter type 4 to cell membranes and improves insulin sensitivity through adenosine monophosphate-activated protein kinase (AMPK) activation, both of which facilitate glucose uptake. Furthermore, 300mg of ALA has been shown to improve endothelial function and reduce fasted blood glucose concentrations in clinical populations. Therefore, investigating the effects of a lower ALA dosage, specifically 200mg, compared to 400mg in the acute fed state, as well as whether ALA and GCE can act synergistically to elicit favourable effects on postprandial glucose control requires further investigation in healthy adults.

Berberine, a known AMPK activator, is a natural alkaloid present in various parts (root, stem, fruit, bark) of multiple plants including, in particular, species found in the Coptis, Hydrastis, and Berberis genus. Chronic berberine supplementation (lasting 1 month) resulted in reduced fasting blood glucose, 2-hour postprandial blood glucose levels, and insulin resistance index scores, outperforming standard care alone in individuals with metabolic syndrome, suggesting that berberine may assist with blood glucose regulation in this population. Berberine has low bioavailability (<1%) reported in both animal and human models largely due to poor intestinal absorption and high levels of first-pass removal in the intestines and liver. To overcome this limitation, higher doses of berberine (500-1500mg) are commonly administered, which may lead to gastrointestinal adverse events. Dihydroberberine (DHB), a highly bioavailable form of berberine, has been shown to achieve greater area under the curve as well as peak berberine concentrations when compared to oral ingestion of 500 mg berberine or placebo in humans. However, whether acute DHB supplementation in combination with green coffee extract elicits beneficial effects on postprandial glucose handling in healthy adults has yet to be elucidated.

The purpose of the current study is to determine the impact of acute supplementation of GCE on postprandial glycemia in healthy adults. A secondary objective is to evaluate the effect of GCE on postprandial insulinemia, insulin sensitivity, glucose oxidation and appetite perceptions. The investigators hypothesize that compared to placebo, a 200mg dose of GCE combined with 400 mg alpha-lipoic acid consumed 30 min prior to a 75g oral glucose challenge will 1) lower 2-hour glucose incremental area under the curve (AUC; primary outcome); 2) lower 2-hour insulin incremental AUC and insulin resistance (Matsuda Index); 3) increase rates of glucose oxidation; and 4) lower appetite perceptions. The investigators also hypothesize that the 200 mg dose of GCE combined with 400 mg alpha-lipoic acid will exert effects like, or greater than, the 200 mg dose of GCE with 200 mg of DHB.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-45 years
* BMI between 18.5-30 kg/m2
* No history of smoking or cardiovascular and metabolic diseases (stroke, hypertension, type II diabetes) or other diseases that could impact the study outcomes
* Weight stable (within ±2kg for 6 months)
* Generally healthy as assessed by medical and physical activity questionnaires
* No oral contraceptive use except for triphasic contraceptives

Exclusion Criteria:

* Any concurrent medical, psychiatric, or orthopedic condition that, subject to investigators' discernment, would negatively affect the subject's ability to comply with the study requirements
* Any history of cardiovascular, neurological, respiratory, skeletal muscle or metabolic disease
* Using medication to manage blood glucose or lipid metabolism
* Bleeding disorders or antiplatelet/ anticoagulation therapy
* Currently using (or use within the last 3 months) monophasic or biphasic oral contraceptives
* Currently supplementing with GCE, ALA, or dihydroberberine
* Any known allergies to green coffee extract, alpha-lipoic acid, dihydroberberine or berberine, or supplementing within the last 3 months
* Currently pregnant or lactating
* Have irregular menstrual cycles (<21 days or >35 days)
* Any form of cancer currently or in the last 5 years
* Are recreational smokers of any form (tobacco or cannabis)
* Use of corticosteroids, testosterone replacement therapy, or any anabolic steroid
* Not willing to consume the 24-hour control diet prior to metabolic trials
* Any current Illness which could interfere with the study (e.g., prolonged diarrhea, regurgitation, etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
2-hour plasma glucose incremental area under the curve | 2 hours
  Determination of the total rise in plasma glucose during an oral glucose tolerance test, to be assessed by an enzyme-linked immunosorbent assay.

SECONDARY OUTCOMES:
2- hour plasma insulin incremental area under the curve | Aggregate 2 hours during the oral glucose tolerance test
  Determination of the total rise in plasma insulin during an oral glucose tolerance test, to be assessed by an enzyme-linked immunosorbent assay.
Postprandial glucose oxidation | Aggregate 2 hours during the oral glucose tolerance test
  Measurement of 13C excretion in breath samples using isotope ratio mass spectrometry.
Appetite perceptions | -30 minutes, 0 minutes, 60 minutes, 120 minutes, during the oral glucose tolerance test.
  "Appetite Visual analog scales" will be used to determine perceptions of hunger, satisfaction, fullness, and prospective food consumption. The maximum values on this scale represent a "Very Strong" appetite perception and the minimum value represents a "Not Strong at All" appetite perception.
Mean glucose concentration | 2 hours
  Mean glucose concentration measured during an oral glucose tolerance test
Mean insulin concentration | 2 hours
  Mean insulin concentration measured during an oral glucose tolerance test
Peak glucose concentration | 2 hours
  Peak glucose concentration measured during an oral glucose tolerance test
Peak insulin concentration | 2 hours
  Peak insulin concentration measured during an oral glucose tolerance test
Insulin sensitivity | 2 hours
  Insulin sensitivity measured via the Matsuda Index during an oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Chris McGlory, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No